CLINICAL TRIAL: NCT04367285
Title: Sensor-based Technology for Upper Limb Rehabilitation in Subject With Multiple Sclerosis: a Randomized Controlled Trial
Brief Title: Sensor-based Technology for Upper Limb Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Marco Tramontano, head of rehabilitation Services, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSLCE/PROG.631
Record Dates: First submitted 2020-04-24; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensor-based Training (Experimental)
  Interventions: Other: Sensor-based Training
- Upper limb motor training (Active Comparator)
  Interventions: Other: Upper limb motor training

INTERVENTIONS:
Other: Sensor-based Training — Sensor-based Training consists of twelve sessions of upper limb training with PABLO®-Tyromotion. For each session the training consists in interactive-games based on virtual reality which allowed a task-oriented approach and a neurocognitive feedback. The exercises require precision tasks and one-dimensional and bidimensional reaction, allowing to train the attention, the strength control and movement control, the coordination and the movement precision. The interactive-games were chosen from those proposed by the Tyromotion PABLO® System.
  Arms: Sensor-based Training
Other: Upper limb motor training — Upper limb motor training, without robotic support. Subjects performed specific exercises aimed to recovery global upper limb functions, to control hand grasp and to improve hand's fine movements.
  Arms: Upper limb motor training

SUMMARY:
Sensor-based technological therapy devices may be good candidates for neuromotor rehabilitation of people with Multiple Sclerosis (MS), especially for treating upper extremities function limitations. The sensor-based device rehabilitation is characterized by interactive therapy games with audio-visual feedback that allows training the movement of shoulders, elbows and wrist, measuring the strength and the active range of motion of upper limb, registering data in an electronic database in order to quantitatively monitoring measures and therapy progress. The aim of this study is to evaluate the effects of sensor-based motor rehabilitation in add-on to the conventional neurorehabilitation, on increasing the upper limbs functions of MS patients. The training consisting of twelve sessions of upper limb training, was compared with twelve sessions of upper limb sensory-motor training, without robotic support. Both rehabilitation programs were performed for 40 minutes three times a week, for 4 weeks, in addition to the conventional therapy. All patients were evaluated at baseline (T0) and after 4 weeks of training (T1)

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Multiple Sclerosis
* upper limb deficits,
* disability between 5 and 8.5 on the Expanded Disability Status Scale (EDSS).

Exclusion Criteria:

* Modified Ashworth Scale (MAS) < 3 at the upper limb;
* cognitive deficits affecting the ability to understand task instructions (Mini-Mental State Examination < 24
* Medical Research Council (MRC) scale with score 0 or 5;
* presence of clinically evaluated severe comorbidities; pregnancy;
* subjects with artificial pacemaker;
* subjects involved in other studies.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in functionality of the upper limb measured in 9 Hole Peg Test (9HPT) at 1 months | 1 month
  Changes in functionality of the upper limb measured in 9-HPT. Changes in the measure in 9-HPT (time, seconds *total scale*) Nine Hole PegTest (Mathiowetz et al, Occup Therap J Resaerach 1985) Time in second to perform the whole test will be recordered (better with less time)

SECONDARY OUTCOMES:
Fatigue Level at 1 month | 1 month
  Fatigue Severity Scale (FSS) is one of the most commonly used self-report questionnaires to measure fatigue. Each question on this scale, which is composed of Likert type questions: 1.I strongly disagree 2.I do not agree 3.No tend to disagree 4. Indefinitely. The total score of the scale, which consists of 9 questions, varies between 9-63. People are asked to mark the appropriate options for each question taking into account their status in the last 1 month period. A total of 36 points and above indicate fatigue
Modified Barthel Index (MBI) at 1 month | 1 month
  Change of Modified Barthel Index (MBI) at 1 month. MBI MBI values ranging from 0 to 105, where 0 means the worse outcome and 105 the best one.
Changes in Multiple Sclerosis Quality of Life-54 questionnaire (MSQOL-54)at 1 month | 1 month
  Change from Baseline in MSQOL-54. MSQOL-54 is a multidimensional health-related quality of life measure, assessing the perception of physical and mental well-being. The instrument is composed of 54 items concerning 12 subscales, which form two scales relating to the physical and mental well-being. The score of the physical function scales, perceptions of health, energy/fatigue, role-physical limitations, pain, sexual function, social function, health distress, is added and corrected to obtain a score on the MSQUOL PHYSICAL HEALTH scale: a score above 50.0 indicates physical well-being. The score of the health distress scale, overall quality of life, emotional well-being, role limitations - emotional, cognitive function is summed and corrected to obtain a score on the scale MSQUOL MENTAL HEALTH: a score above 50.0 indicates mental well-being. The administration time is about 11-18 minutes, it can be completed by an interviewer or by the patient.
Changes of Medical Research Council scale (MRC) at 1 month | 1 month
  The MRC score is obtained by evaluating 12 muscle groups in the upper extremities (wrist extensors, elbow flexors and abductors of the shoulder) and lower extremities (dorsal ankle flexors, knee extensors, and hip flexors). For each muscle group will be assigned a score between 0 (complete paralysis) and 5 (normal force), and the total score can vary between 0 up to 60 points.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Tramontano, Principal Investigator — SANTA LUCIA FOUNDATION
Locations (1):
- Marco Tramontano, Rome, Italy

IPD SHARING:
Plan to Share IPD: No